CLINICAL TRIAL: NCT02772081
Title: An Open-Label, Multicenter, Randomized, Controlled Study in Spontaneously Breathing Preterm Neonates With Respiratory Distress Syndrome to Compare Two Procedures for Porcine Surfactant (Poractant Alfa, CUROSURF®) Administration: A Less Invasive Method (LISA) During Non-invasive Ventilation (NIV) and the Conventional Administration During Brief Invasive Ventilation.
Brief Title: A Study in Preterm Neonates With Respiratory Distress Syndrome (RDS) Comparing CUROSURF® Administration Through Less Invasive Surfactant Administration (LISA) and Conventional Administration
Acronym: LISPAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-050000-01
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Distress Syndrome (RDS)
Keywords: Less Invasive Surfactant administration; LISPAP; Neonates; Newborns; Respiratory Distress Syndrome (RDS); CUROSURF®
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Curosurf LISA (Experimental): Single dose of poractant alfa 200 mg/kg via brief insertion of a thin catheter (CHF 6440) into the trachea in neonates with RDS.
  A second surfactant dose at 100 mg/kg will be administered with the same technique as the first dosage administration if needed.
  After the first and second surfactant administration, neonates could receive a third surfactant dose at 100 mg/kg through a standard technique if needed.
  Interventions: Combination Product: LISA combination product (Curosurf+catheter CHF6440)
- Curosurf Endotracheal Tube (Active Comparator): Single dose of poractant alfa 200 mg/kg via the conventional intubation with endotracheal tube in neonates with RDS.
  A second surfactant dose at 100 mg/kg will be administered with the same technique as the first dosage administration if needed.
  After the first and second surfactant administration, neonates could receive a third surfactant dose at 100 mg/kg through a standard technique if needed.
  Interventions: Drug: Curosurf through conventional administration (endotracheal tube)

INTERVENTIONS:
Combination Product: LISA combination product (Curosurf+catheter CHF6440) — Curosurf administration through brief insertion of a thin catheter into the trachea
  Arms: Curosurf LISA
Drug: Curosurf through conventional administration (endotracheal tube) — Curosurf through conventional administration (endotracheal tube), followed by rapid extubation
  Arms: Curosurf Endotracheal Tube

SUMMARY:
This study compared the administration of porcine surfactant (poractant alfa, Curosurf®) through a less invasive method (LISA), using a thin catheter, CHF 6440 (LISACATH®), during non-invasive ventilation (CPAP, NIPPV, BiPAP) with an approved conventional surfactant administration during invasive ventilation followed by rapid extubation in terms of short term and mid-term safety and efficacy in spontaneously breathing preterm neonates who have clinical signs of respiratory distress syndrome (RDS).

DETAILED DESCRIPTION:
This study was an open-label, multicentre, randomized, controlled study of spontaneously breathing neonates with RDS. Neonates were evaluated according to the selection criteria and then randomized to surfactant treatment via LISA or standard administration procedure. The enrolment was staggered: the gestational age was restricted to 27+0 weeks up to 28+6 weeks for the first 15 neonates. Provided no safety concerns were raised, the enrolment was planned to be extended to the whole population (i.e. 25+0 weeks up to 28+6 weeks). Enrolled neonates were evaluated in a main phase of the trial until discharge or 40 weeks post-menstrual age (PMA), whichever came first. Their clinical status and neurodevelopment was to be assessed at 24-month corrected age as a separate stand-alone visit.

The Sponsor decided to terminate the study early, due to uncertain sufficient availability of the CHF 6440 catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained by parents/legal representative (according to local regulation) prior to or after birth
2. Preterm neonates of either sex aged ≥30 minutes and <24 hours, spontaneously breathing and stabilized on non-invasive ventilation (NIV).
3. Gestational age of 25+0 weeks up to 28+6 completed weeks, except for the first 15 enrolled neonates in which the gestational age will be restricted to 27+0 weeks up to 28+6 weeks.
4. Clinical course consistent with RDS.
5. Fraction of inspired oxygen (FiO2) ≥0.30 to maintain preductal oxygen saturation (SpO2) between 88-95%.

Exclusion Criteria:

1. Need for immediate endotracheal intubation for cardiopulmonary resuscitation or insufficient respiratory drive
2. Use of nasal high frequency oscillatory ventilation (nHFOV) prior to study entry
3. Use of surfactant prior to study entry and need for intratracheal administration of any other treatment (e.g. nitric oxide)
4. Known genetic or chromosomal disorders, major congenital anomalies (congenital heart diseases, myelomeningocele etc)
5. Mothers with prolonged rupture of the membranes (> 21 days duration)
6. Presence of air leaks if identified and known prior to study entry
7. Evidence of severe birth asphyxia (e.g. continued need for resuscitation at 10 minutes after birth, altered neurological state, or neonatal encephalopathy)
8. Neonatal seizures prior to study entry
9. Any condition that, in the opinion of the Investigator, would place the neonate at undue risk
10. Participation in another clinical trial of any medicinal product, placebo, experimental medical device, or biological substance conducted under the provisions of a protocol on the same therapeutic target.

Ages: 30 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rangasamy Ramanathan, M.D., Principal Investigator — LAC+USC Medical Center & Good Samaritan Hospital
Locations (26):
- United States (26):
  - Chiesi Clinical Trial Site 84029, Little Rock, Arkansas
  - Chiesi Clinical Trial Site 84001, Los Angeles, California
  - Chiesi Clinical Trial Site 84002, Los Angeles, California
  - Chiesi Clinical Trial Site 84013, Denver, Colorado
  - Chiesi Clinical Trial Site 84026, New Britain, Connecticut
  - Chiesi Clinical Trial Site 84003, Evanston, Illinois
  - Chiesi Clinical Trial Site 84021, Peoria, Illinois
  - Chiesi Clinical Trial Site 84023, Lexington, Kentucky
  - Chiesi Clinical Trial Site 84028, Springfield, Massachusetts
  - Chiesi Clinical Trial Site 84005, Worcester, Massachusetts
  - Chiesi Clinical Trial Site 84008, Lansing, Michigan
  - Chiesi Clinical Trial Site 84004, St Louis, Missouri
  - Chiesi Clinical Trial Site 84012, Camden, New Jersey
  - Chiesi Clinical Trial Site 84024, Manhasset, New York
  - Chiesi Clinical Trial Site 84019, New Hyde Park, New York
  - Chiesi Clinical Trial Site 84009, Valhalla, New York
  - Chiesi Clinical Trial Site 84027, Greenville, North Carolina
  - Chiesi Clinical Trial Site 84010, Wilmington, North Carolina
  - Chiesi Clinical Trial Site 84025, Cincinnati, Ohio
  - Chiesi Clinical Trial Site 84017, Oklahoma City, Oklahoma
  - Chiesi Clinical Trial Site 84020, Hershey, Pennsylvania
  - Chiesi Clinical Trial Site 84007, Nashville, Tennessee
  - Chiesi Clinical Trial Site 84011, Lubbock, Texas
  - Chiesi Clinical Trial Site 84006, Plano, Texas
  - Chiesi Clinical Trial Site 84022, Temple, Texas
  - Chiesi Clinical Trial Site 84015, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-001974-14/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Curosurf LISA: Single dose of poractant alfa 200 mg/kg via brief insertion of a thin catheter (CHF 6440) into the trachea in neonates with RDS.
  A second surfactant dose at 100 mg/kg will be administered with the same technique as the first dosage administration if needed.
  After the first and second surfactant administration, neonates could receive a third surfactant dose at 100 mg/kg through a standard technique if needed.
  LISA combination product (Curosurf+catheter CHF6440): Curosurf administration through brief insertion of a thin catheter into the trachea
- Curosurf Endotracheal Tube: Single dose of poractant alfa 200 mg/kg via the conventional intubation with endotracheal tube in neonates with RDS.
  A second surfactant dose at 100 mg/kg will be administered with the same technique as the first dosage administration if needed.
  After the first and second surfactant administration, neonates could receive a third surfactant dose at 100 mg/kg through a standard technique if needed.
  Curosurf through conventional administration (endotracheal tube): Curosurf through conventional administration (endotracheal tube), followed by rapid extubation
Period: Overall Study
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Started | 20 | 13
Completed | 18 | 11
Not Completed | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube | Total
Number analyzed (Participants) | 19 | 12 | 31
Age, Continuous [Mean (Full Range); unit: weeks] — Gestational age at birth.
  weeks | 27.65 [26.3 to 28.9] | 27.92 [26.3 to 28.9] | 27.76 [26.3 to 28.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants] — Population: Neonate and maternal demographic and baseline characteristics are based on the ITT population
  participants
    Hispanic or Latino | 5 | 6 | 11
    Not Hispanic or Latino | 14 | 6 | 20
Region of Enrollment [Number; unit: participants]
  United States | 19 | 12 | 31
Birth weight [Mean (Full Range); unit: kg] | 1.009 [0.56 to 1.67] | 0.973 [0.52 to 1.64] | 0.995 [0.52 to 1.67]
APGAR score at 1 minute post-birth [Mean (Full Range); unit: scores on a scale] — The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7 to 10 is normal and is a sign that the newborn is in good health. A baby who scores under a 7 may require immediate medical care.
  scores on a scale | 5.6 [2 to 8] | 4.8 [2 to 6] | 5.3 [2 to 8]
APGAR score at 5 minutes post-birth [Mean (Full Range); unit: APGAR score] — The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7 to 10 is normal and is a sign that the newborn is in good health. A baby who scores under a 7 may require immediate medical care.
  APGAR score | 7.5 [5 to 9] | 7.7 [6 to 9] | 7.6 [5 to 9]
Mother's age [Mean (Full Range); unit: years] | 30.0 [22.0 to 39.0] | 25.8 [18.0 to 34.0] | 28.4 [18 to 39]
Mother's race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 11 | 8 | 19
  Unknown or Not Reported | 2 | 1 | 3
Mother's ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 13 | 5 | 18
  Data missing | 1 | 1 | 2
Antibiotics taken - YES [Count of Participants; unit: Participants] | 9 | 8 | 17
Corticosteroids taken -- YES [Count of Participants; unit: Participants] | 14 | 11 | 25
Number of days from last corticosteroid dose up to birth, [Number; unit: days] — Population: The information refers to the mothers of enrolled subjects, who took antibiotics and corticosteroids during pregnancy.
  days
    0-1 days: number analyzed (Participants) | 14 | 11 | 25
    0-1 days | 8 | 5 | 13
    2-7 days: number analyzed (Participants) | 14 | 11 | 25
    2-7 days | 3 | 6 | 9
    >7 days: number analyzed (Participants) | 14 | 11 | 25
    >7 days | 3 | 0 | 3
Type of delivery [Count of Participants; unit: Participants]
  C-section with labor | 2 | 3 | 5
  C-section without labor | 10 | 4 | 14
  Emergency C-section | 5 | 3 | 8
  Spontaneous | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety: Study Treatment Administration: Number of Participants Who Received 1, 2, or 3 Doses of Treatment
Description: Extent of exposure to study treatment is summarized by treatment group. Number of participants who received 1, 2, or 3 doses of treatment.
  All neonates received the first administration of Curosurf® 200 mg/kg. In case of lack of efficacy or clinical deterioration, a second dose of Curosurf® 100 mg/kg was administered using the same technique as the first dose. Neonates could receive a third Curosurf® 100 mg/kg dose if needed, administered using a standard technique. Results are presented as the number of neonates who received 1, 2, or 3 doses of Curosurf®, administered.
Time Frame: First 72 hours of life.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
Participants
  Number of Curosurf® dose, n=1 dose | 13 | 9
  Number of Curosurf® doses, n=2 doses | 4 | 2
  Number of Curosurf® doses, n=3 doses | 2 | 1

2. Primary Outcome: Safety: Study Treatment Administration: Number of Participants for Whom the First Attempt Failed to Insert the Catheter/Endotracheal Tube
Description: Number of participants for whom the first attempt failed to insert the catheter/endotracheal tube and the percentage of neonates with first failed attempt, is presented by treatment group.
Time Frame: At first surfactant administration, up to Day 1.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
Participants | 5 | 5
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; First Administration; Treatment comparison. Adjusted difference, its 95% confidence interval (CI) and p-value are estimated using Cochran-Mantel-Haenszel test; Test type: Superiority; p = 0.390, Cochran-Mantel-Haenszel; Adjusted difference = -15.4, 95% CI 2-sided [-47.9 to 17.1]

3. Primary Outcome: Safety: Study Treatment Administration: Number of Maneuvers Discontinued Due to Neonate's Severe Destabilization
Description: Number of manoeuvres (attempts) discontinued, due to neonate's severe destabilization is presented by treatment group.
Time Frame: At first surfactant administration, up to Day 1 or at second administration, up to 2 days.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: Number of maneuvers (attempts)
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
Number of maneuvers (attempts)
  First administration: number analyzed (Participants) | 18 | 12
  First administration | 0.1 [0 to 1] | 0.0 [0 to 0]
  Second administration: number analyzed (Participants) | 4 | 3
  Second administration | 0.3 [0 to 1] | 0.0 [0 to 0]

4. Primary Outcome: Safety: Study Treatment Administration: Number of Attempts to First Successful Insertion
Description: Number of attempts required to achieve first successful insertion is presented by treatment group.
Time Frame: At first surfactant administration, up to Day 1 or at second administration, up to 2 days.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: Number of maneuvers (attempts)
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
Number of maneuvers (attempts)
  First administration | 1.3 [1 to 2] | 1.8 [1 to 5]
  Second administration: number analyzed (Participants) | 4 | 2
  Second administration | 2.0 [1 to 3] | 1.0 [1 to 1]

5. Primary Outcome: Safety: Study Treatment Administration: Number of Device Misallocation for LISA Administration Group (Esophageal Insertion)
Description: Number of device misallocation for LISA administration group (esophageal insertion).
  Data was not collected from participants in the "Curosurf Endotracheal Tube" -- the control arm of the study, because it is not applicable.
Time Frame: At first surfactant administration, up to Day 1 or at second administration, up to 2 days.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: Number of maneuvers (attempts)
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 0
Number of maneuvers (attempts)
  First administration | 0.2 [0 to 1] |
  Second administration | 0.0 [0 to 0] |

6. Primary Outcome: Safety: Study Treatment Administration: Duration of Surfactant Administration
Description: Duration of surfactant administration is presented by treatment group.
Time Frame: At first surfactant administration, up to Day 1 or at second administration, up to 2 days.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
minutes
  First administration | 1.8 [1 to 5] | 2.3 [1 to 4]
  Second administration: number analyzed (Participants) | 4 | 3
  Second administration | 2.3 [1 to 4] | 1.7 [0 to 3]

7. Primary Outcome: Safety: Study Treatment Administration: Duration of the Whole Procedure
Description: Duration of the whole procedure (starting from the insertion of laryngoscope up to the removal of the catheter/ETT), is presented by treatment group.
Time Frame: At first surfactant administration, up to Day 1 or at second administration, up to 2 days.
Population: Safety population (SAF): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
minutes
  First administration: number analyzed (Participants) | 19 | 11
  First administration | 3.9 [1 to 10] | 7.8 [2 to 15]
  Second administration: number analyzed (Participants) | 4 | 1
  Second administration | 5.8 [2 to 10] | 3.0 [3 to 3]

8. Secondary Outcome: Efficacy: Duration of Oxygen Alone Supplementation and Any Non-Invasive Ventilation (NIV)
Description: The duration of oxygen alone supplementation and any non-invasive ventilation (NIV) during the study are presented by treatment group.
  PMA=Post-Menstrual Age PNA=Post-Natal Age
Time Frame: First 72 hours of life, Up to 28 days Post-Natal Age (PNA), Up to 36 weeks Post-Menstrual Age (PMA).
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: days
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
days
  Duration of standalone oxygen supplementation: number analyzed (Participants) | 9 | 8
  Duration of standalone oxygen supplementation | 16.4 [3 to 27] | 16.4 [3 to 52]
  Duration of NIV | 45.7 [2 to 87] | 38.3 [1 to 70]
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Duration of standalone oxygen supplementation; Test type: Superiority; p = 0.563, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 5.0, 95% CI 2-sided [-13.8 to 23.8]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Duration of NIV; Test type: Superiority; p = 0.612, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [-19.7 to 21.7]

9. Secondary Outcome: Efficacy: Neonates Needing Additional 2 or 3 Doses of Surfactant
Description: A summary of the percentage of neonates requiring at least one additional dose of surfactant, and respective statistical analysis, is presented by treatment group i.e. 2 or 3 doses of surfactant .
Time Frame: First 72 hours of life.
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 6 | 3
Participants
  Additional dose of surfactant (n=2 doses) | 4 | 2
  Additional dose of surfactant (n=3 doses) | 2 | 1

10. Secondary Outcome: Efficacy: Neonates Needing Additional Surfactant Doses
Description: A summary of the percentage of neonates requiring at least one additional dose of surfactant, and respective statistical analysis, is presented by treatment group.
Time Frame: First 72 hours of life.
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
Participants | 6 | 3

11. Secondary Outcome: Efficacy: Preductal Oxygen Saturation/Fraction of Inspired Oxygen (SpO2/FiO2) Ratio
Description: The mean SpO2/FiO2 ratio values at timepoints up to and including 120 hours post-treatment, and respective statistical analyses, are summarized by treatment group.
Time Frame: Pre-procedure, at time 0 (T0, end of surfactant instillation) and post treatment after T0 at 5, 15, 30 minutes, at 1, 6, 12, 24, 48, 72, and 120 hours, on Day 28 PNA, 36 weeks PMA.
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
ratio
  Pre-procedure | 2.368 (0.794) | 2.052 (0.659)
  T0: number analyzed (Participants) | 19 | 10
  T0 | 1.796 (1.035) | 2.463 (1.221)
  5 mins: number analyzed (Participants) | 19 | 10
  5 mins | 3.113 (1.164) | 2.657 (1.376)
  15 mins: number analyzed (Participants) | 18 | 10
  15 mins | 3.438 (1.116) | 3.010 (1.229)
  30 mins | 3.960 (0.875) | 3.253 (1.358)
  1 hour | 4.106 (0.869) | 3.577 (0.921)
  6 hours | 4.152 (0.776) | 3.919 (1.061)
  12 hours | 4.090 (0.811) | 3.976 (1.172)
  24 hours | 4.139 (0.730) | 3.829 (0.945)
  48 hours: number analyzed (Participants) | 19 | 11
  48 hours | 4.046 (0.568) | 3.653 (0.952)
  72 hours: number analyzed (Participants) | 19 | 11
  72 hours | 3.988 (0.887) | 3.916 (0.944)
  120 hours: number analyzed (Participants) | 19 | 11
  120 hours | 4.205 (0.698) | 4.263 (0.862)
  Day 28 PNA: number analyzed (Participants) | 18 | 11
  Day 28 PNA | 3.975 (1.104) | 3.804 (0.936)
  36 weeks PMA: number analyzed (Participants) | 4 | 4
  36 weeks PMA | 3.571 (0.535) | 3.840 (0.599)
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; T0, Treatment comparison. The analysis was based on an mixed model for repeated measures (MMRM) with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.137, Mixed model for repeated measures; Adjusted mean difference = -0.619, 95% CI 2-sided [-1.447 to 0.210]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 5 min, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.534, Mixed model for repeated measures; Adjusted mean difference = 0.268, 95% CI 2-sided [-0.604 to 1.140]
Statistical Analysis 3: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 15 min, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.530, Mixed model for repeated measures; Adjusted mean difference = 0.270, 95% CI 2-sided [-0.597 to 1.136]
Statistical Analysis 4: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 30 min, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.091, Mixed model for repeated measures; Adjusted mean difference = 0.641, 95% CI 2-sided [-0.108 to 1.389]
Statistical Analysis 5: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 1 hour, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.040, Mixed model for repeated measures; Adjusted mean difference = 0.463, 95% CI 2-sided [0.023 to 0.903]
Statistical Analysis 6: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 6 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.532, Mixed model for repeated measures; Adjusted mean difference = 0.166, 95% CI 2-sided [-0.371 to 0.703]
Statistical Analysis 7: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 12 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.877, Mixed model for repeated measures; Adjusted mean difference = 0.048, 95% CI 2-sided [-0.578 to 0.674]
Statistical Analysis 8: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 24 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.356, Mixed model for repeated measures; Adjusted mean difference = 0.244, 95% CI 2-sided [-0.289 to 0.776]
Statistical Analysis 9: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 48 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.258, Mixed model for repeated measures; Adjusted mean difference = 0.303, 95% CI 2-sided [-0.235 to 0.841]
Statistical Analysis 10: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 72 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.945, Mixed model for repeated measures; Adjusted mean difference = 0.022, 95% CI 2-sided [-0.616 to 0.660]
Statistical Analysis 11: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 120 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2/FiO2 as a covariate; Test type: Superiority; p = 0.766, Mixed model for repeated measures; Adjusted mean difference = -0.075, 95% CI 2-sided [-0.586 to 0.436]

12. Secondary Outcome: Efficacy: Fraction of Inspired Oxygen (FiO2)
Description: The FiO2 values at timepoints up to and including 120 hours post-treatment and the changes from pre-procedure to each of those timepoints are presented by treatment group.
  The fraction of inspired oxygen (FiO2) is the concentration of oxygen in the gas mixture.
Time Frame: as for outcome 11
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: fraction of inspired oxygen
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
fraction of inspired oxygen
  Pre-procedure | 0.435 (0.151) | 0.524 (0.235)
  T0: number analyzed (Participants) | 19 | 10
  T0 | 0.569 (0.252) | 0.475 (0.250)
  5 mins: number analyzed (Participants) | 19 | 10
  5 mins | 0.365 (0.197) | 0.457 (0.260)
  15 mins: number analyzed (Participants) | 18 | 10
  15 mins | 0.321 (0.199) | 0.373 (0.186)
  30 mins | 0.257 (0.090) | 0.372 (0.258)
  1 hour | 0.251 (0.108) | 0.279 (0.084)
  6 hours | 0.244 (0.077) | 0.274 (0.131)
  12 hours | 0.246 (0.075) | 0.290 (0.225)
  24 hours | 0.238 (0.064) | 0.269 (0.113)
  48 hours: number analyzed (Participants) | 19 | 11
  48 hours | 0.239 (0.033) | 0.285 (0.133)
  72 hours: number analyzed (Participants) | 19 | 11
  72 hours | 0.257 (0.088) | 0.262 (0.099)
  120 hours: number analyzed (Participants) | 19 | 11
  120 hours | 0.237 (0.049) | 0.243 (0.099)
  Day 28 PNA: number analyzed (Participants) | 18 | 11
  Day 28 PNA | 0.285 (0.188) | 0.272 (0.091)
  36 weeks PMA: number analyzed (Participants) | 4 | 5
  36 weeks PMA | 0.270 (0.029) | 0.254 (0.033)
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; T0, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.590, Mixed model for repeated measures; Adjusted mean difference = 0.051, 95% CI 2-sided [-0.141 to 0.243]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 5 min, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.511, Mixed model for repeated measures; Adjusted mean difference = -0.051, 95% CI 2-sided [-0.210 to 0.107]
Statistical Analysis 3: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 15 min, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.488, Mixed model for repeated measures; Adjusted mean difference = -0.050, 95% CI 2-sided [-0.196 to 0.096]
Statistical Analysis 4: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 30 min, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.091, Mixed model for repeated measures; Adjusted mean difference = -0.110, 95% CI 2-sided [-0.239 to 0.019]
Statistical Analysis 5: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 1 hour, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.344, Mixed model for repeated measures; Adjusted mean difference = -0.024, 95% CI 2-sided [-0.076 to 0.027]
Statistical Analysis 6: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 6 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.376, Mixed model for repeated measures; Adjusted mean difference = -0.026, 95% CI 2-sided [-0.084 to 0.033]
Statistical Analysis 7: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 12 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.396, Mixed model for repeated measures; Adjusted mean difference = -0.040, 95% CI 2-sided [-0.135 to 0.055]
Statistical Analysis 8: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 24 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.268, Mixed model for repeated measures; Adjusted mean difference = -0.026, 95% CI 2-sided [-0.074 to 0.021]
Statistical Analysis 9: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 48 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.147, Mixed model for repeated measures; Adjusted mean difference = -0.037, 95% CI 2-sided [-0.089 to 0.014]
Statistical Analysis 10: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 72 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.994, Mixed model for repeated measures; Adjusted mean difference = 0.000, 95% CI 2-sided [-0.055 to 0.055]
Statistical Analysis 11: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 120 hours, Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure FiO2 as a covariate; Test type: Superiority; p = 0.853, Mixed model for repeated measures; Adjusted mean difference = -0.004, 95% CI 2-sided [-0.048 to 0.040]

13. Secondary Outcome: Efficacy: Preductal Oxygen Saturation (SpO2)
Description: The mean SpO2 values at timepoints up to and including 120 hours post-treatment are summarized by treatment group.
  Oxygen saturation (SpO2) is a measurement of how much oxygen the blood is carrying as a percentage of the maximum it could carry.
Time Frame: as for outcome 11
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
percentage of oxygen saturation
  Pre-procedure | 92.7 (3.0) | 94.3 (3.4)
  T0: number analyzed (Participants) | 19 | 10
  T0 | 81.1 (17.9) | 93.3 (6.6)
  5 mins: number analyzed (Participants) | 19 | 10
  5 mins | 94.6 (7.6) | 93.7 (7.1)
  15 mins: number analyzed (Participants) | 18 | 10
  15 mins | 92.8 (9.6) | 93.5 (4.7)
  30 mins | 95.0 (4.1) | 91.3 (10.6)
  1 hour | 94.5 (4.8) | 93.0 (3.7)
  6 hours | 96.1 (2.6) | 94.8 (2.7)
  12 hours | 94.9 (3.1) | 91.9 (14.0)
  24 hours | 94.5 (3.6) | 93.9 (4.5)
  48 hours: number analyzed (Participants) | 19 | 11
  48 hours | 95.2 (2.9) | 93.6 (2.9)
  72 hours | 95.5 (2.9) | 93.8 (3.6)
  120 hours | 96.4 (2.7) | 95.6 (2.2)
  Day 28 PNA: number analyzed (Participants) | 18 | 11
  Day 28 PNA | 96.3 (3.4) | 96.0 (2.9)
  36 weeks PMA: number analyzed (Participants) | 8 | 7
  36 weeks PMA | 97.0 (3.3) | 96.6 (2.1)
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; T0; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.090, Mixed model for repeated measures; Adjusted mean difference = -10.4, 95% CI 2-sided [-22.6 to 1.7]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 5 min; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.917, Mixed model for repeated measures; Adjusted mean difference = -0.3, 95% CI 2-sided [-6.4 to 5.8]
Statistical Analysis 3: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 15 min; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.668, Mixed model for repeated measures; Adjusted mean difference = -1.5, 95% CI 2-sided [-8.5 to 5.6]
Statistical Analysis 4: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 30 min; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.149, Mixed model for repeated measures; Adjusted mean difference = 4.0, 95% CI 2-sided [-1.5 to 9.6]
Statistical Analysis 5: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 1 hour; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.318, Mixed model for repeated measures; Adjusted mean difference = 1.8, 95% CI 2-sided [-1.9 to 5.5]
Statistical Analysis 6: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 6 hour; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.148, Wilcoxon (Mann-Whitney); Adjusted mean difference = 1.6, 95% CI 2-sided [-0.6 to 3.7]
Statistical Analysis 7: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 12 hours; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.333, Mixed model for repeated measures; Adjusted mean difference = 3.3, 95% CI 2-sided [-3.6 to 10.2]
Statistical Analysis 8: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 24 hours; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.560, Mixed model for repeated measures; Adjusted mean difference = 0.9, 95% CI 2-sided [-2.2 to 4.0]
Statistical Analysis 9: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 48 hours; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.089, Mixed model for repeated measures; Adjusted mean difference = 2.0, 95% CI 2-sided [-0.3 to 4.3]
Statistical Analysis 10: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 72 hours; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.115, Mixed model for repeated measures; Adjusted mean difference = 1.9, 95% CI 2-sided [-0.5 to 4.4]
Statistical Analysis 11: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; 120 hours; Treatment comparison. The analysis was based on an MMRM with treatment, timepoint, treatment by timepoint interaction, and GA group as fixed effects and pre-procedure SpO2 as a covariate; Test type: Superiority; p = 0.284, Mixed model for repeated measures; Adjusted mean difference = 1.1, 95% CI 2-sided [-1.0 to 3.3]

14. Secondary Outcome: Efficacy: Percentage of Neonates Needing Any Intubation Procedure, Outside the Initial Surfactant Administration Period
Description: The percentage of neonates needing any intubation procedure, outside the initial surfactant administration period (i.e., excluding endotracheal intubation[s] that were required for surfactant administration in the Conventional administration arm), in the first 72 hours of life, in the first 28 days post-natal age (PNA), and within 36 weeks Post-menstrual age (PMA), and respective statistical analyses, are presented.
Time Frame: First 72 hours of life, up to 28 days post-natal age (PNA), Up to 36 weeks Post-menstrual age (PMA)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
percentage of participants
  Any intubation procedure in first 72 hours of life. | 10.5 | 25.0
  Any intubation procedure in first 28 days PNA | 31.6 | 25.0
  Any intubation procedure within 36 weeks PMA | 31.6 | 25.0
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Any intubation procedure in first 72 hours of life; Test type: Superiority; p = 0.220, Cochran-Mantel-Haenszel; Adjusted difference = -15.7, 95% CI 2-sided [-39.6 to 8.2]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Any intubation procedure within 36 weeks PMA; Test type: Superiority; p = 0.741, Cochran-Mantel-Haenszel; Adjusted difference = 4.9, 95% CI 2-sided [-22.8 to 32.5]

15. Secondary Outcome: Efficacy: Median Duration of Invasive Mechanical Ventilation During the Study
Description: The duration of invasive ventilation (MV) in the first 28 days PNA, and within 36 weeks PMA, are presented by treatment group.
  Participants who actually received invasive ventilation are reported in the table below.
Time Frame: Up to 28 days PNA, Up to 36 weeks PMA
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
days
  Duration of invasive MV in first 28 days PNA: number analyzed (Participants) | 6 | 4
  Duration of invasive MV in first 28 days PNA | 6.0 [4 to 18] | 20.5 [2 to 27]
  Duration of invasive MV within 36 weeks PMA: number analyzed (Participants) | 6 | 4
  Duration of invasive MV within 36 weeks PMA | 6 [4 to 18] | 24 [2 to 45]
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Duration of invasive MV in first 28 days PNA; Test type: Superiority; p = 0.333, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -8.0, 95% CI 2-sided [-32.3 to 16.3]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Duration of invasive MV within 36 weeks PMA; Test type: Superiority; p = 0.334, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -8.0, 95% CI 2-sided [-49.5 to 33.5]

16. Secondary Outcome: Efficacy: Duration of Invasive Mechanical Ventilation During the Study
Description: The duration of invasive ventilation (MV) in the first 72 hours of life and respective statistical analyses, are presented by treatment group.
Time Frame: First 72 hours of life
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Median (Full Range); unit: hours
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 3 | 4
hours | 29.8 [6 to 67] | 61.4 [19 to 68]
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Duration of invasive mechanical ventilation; Test type: Superiority; p = 0.596, Wilcoxon (Mann-Whitney); Adjusted difference = -28.6, 95% CI 2-sided [-120.9 to 63.6]

17. Secondary Outcome: Efficacy: Percentage of Neonates Needing Invasive Mechanical Ventilation (MV) During the Study
Description: The percentage of neonates needing invasive mechanical ventilation (MV) in the first 72 hours of life, in the first 28 days post-natal age (PNA), and within 36 weeks Post-Menstrual Age (PMA), and respective statistical analyses, are presented by treatment group.
Time Frame: First 72 hours of life, Up to 28 days Post-Natal Age (PNA), Up to 36 weeks PMA
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
Participants
  Invasive MV in first 72 hours of life. | 3 | 4
  Invasive MV in first 28 days PNA. | 6 | 4
  Invasive MV within 36 weeks PMA. | 6 | 4
Statistical Analysis 1: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Invasive MV in the first 72 hours of life; Test type: Superiority; p = 0.219, Cochran-Mantel-Haenszel — The percentage of neonates needing invasive MV in the first 72 hours of life, was compared between the treatment groups using the Cochran-Mantel-Haenszel (CMH) test, adjusted for gestational age (GA) group; CMH adjusted difference = -18.6, 95% CI 2-sided [-47.0 to 9.8]
Statistical Analysis 2: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Invasive MV in first 28 days PNA; Test type: Superiority; p = 0.826, Cochran-Mantel-Haenszel; Adjusted difference = -3.4, 95% CI 2-sided [-33.5 to 26.7]
Statistical Analysis 3: Comparison: Curosurf LISA vs Curosurf Endotracheal Tube; Invasive MV within 36 weeks PMA; Test type: Superiority; p = 0.826, Cochran-Mantel-Haenszel; Adjusted difference = -3.4, 95% CI 2-sided [-33.5 to 26.7]

18. Secondary Outcome: Efficacy: Blood Gas Analysis Parameters -- pH
Description: The blood gas analysis for blood pH at all timepoints and the changes from pre-procedure to each timepoint are presented.
  Results for pH values are based on a scale of 0 to 14. A pH value of 7 is neutral, pH less than 7 is acidic, and pH greater than 7 is basic.
Time Frame: First 72 hours of life (1h, 6h, 24h, 48h, 72h)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: units on a pH scale
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
units on a pH scale
  Pre-procedure (actual value): number analyzed (Participants) | 18 | 11
  Pre-procedure (actual value) | 7.289 [7.21 to 7.37] | 7.240 [7.05 to 7.34]
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure): number analyzed (Participants) | 17 | 10
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure) | 0.016 [-0.07 to 0.07] | 0.038 [-0.04 to 0.15]
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure): number analyzed (Participants) | 17 | 10
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure) | 0.044 [-0.04 to 0.13] | 0.047 [-0.05 to 0.19]
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure): number analyzed (Participants) | 17 | 10
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure) | 0.038 [-0.05 to 0.22] | 0.082 [-0.06 to 0.25]
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure): number analyzed (Participants) | 16 | 9
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure) | 0.008 [-0.11 to 0.12] | 0.072 [-0.08 to 0.19]
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure): number analyzed (Participants) | 17 | 9
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure) | 0.001 [-0.16 to 0.14] | 0.068 [-0.04 to 0.14]

19. Secondary Outcome: Efficacy: Blood Gas Analysis Parameters -- Partial Pressure of Carbon Dioxide (pCO2)
Description: The blood gas analysis partial pressure of carbon dioxide (pCO2) at all timepoints and the changes from pre-procedure to each timepoint are presented.
Time Frame: First 72 hours of life (1h, 6h, 24h, 48h, 72h)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
mmHg
  Pre-procedure (actual value): number analyzed (Participants) | 18 | 11
  Pre-procedure (actual value) | 50.30 [39.2 to 67.0] | 52.34 [24.0 to 93.0]
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure): number analyzed (Participants) | 17 | 10
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure) | -4.00 [-16.0 to 6.0] | -0.85 [-18.0 to 8.0]
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure): number analyzed (Participants) | 17 | 10
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure) | -7.55 [-27.0 to 3.0] | -2.26 [-35.0 to 11.0]
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure): number analyzed (Participants) | 17 | 10
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure) | -6.12 [-35.0 to 5.0] | -7.93 [-45.0 to 18.0]
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure): number analyzed (Participants) | 16 | 9
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure) | -2.70 [-22.0 to 25.0] | -5.64 [-31.0 to 18.0]
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure): number analyzed (Participants) | 17 | 9
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure) | -2.92 [-24.0 to 19.0] | -5.24 [-26.2 to 15.0]

20. Secondary Outcome: Efficacy: Blood Gas Analysis Parameters -- Partial Pressure of Oxygen (pO2)
Description: The blood gas analysis partial pressure of oxygen (pO2) at all timepoints and the changes from pre-procedure to each timepoint are presented.
Time Frame: First 72 hours of life (1h, 6h, 24h, 48h, 72h)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
mmHg
  Pre-procedure (actual value): number analyzed (Participants) | 18 | 11
  Pre-procedure (actual value) | 54.78 [20.0 to 88.0] | 58.51 [10.0 to 91.0]
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure): number analyzed (Participants) | 17 | 10
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure) | 4.22 [-32.0 to 69.0] | 2.34 [-31.0 to 68.0]
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure): number analyzed (Participants) | 17 | 10
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure) | 2.69 [-31.0 to 27.0] | -0.06 [-67.0 to 63.0]
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure): number analyzed (Participants) | 17 | 10
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure) | -5.74 [-52.0 to 27.0] | 0.84 [-34.0 to 54.0]
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure): number analyzed (Participants) | 16 | 9
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure) | -7.51 [-37.0 to 33.0] | -8.07 [-54.0 to 29.0]
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure): number analyzed (Participants) | 17 | 8
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure) | -5.01 [-34.1 to 52.0] | -2.25 [-40.0 to 51.0]

21. Secondary Outcome: Efficacy: Blood Analysis Parameter -- Bicarbonate (HCO3^-)
Description: The blood concentration of bicarbonate (HCO3^-) at all timepoints and the changes from pre-procedure to each timepoint are presented.
Time Frame: First 72 hours of life (1h, 6h, 24h, 48h, 72h)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
mmol/L
  Pre-procedure (actual value): number analyzed (Participants) | 18 | 11
  Pre-procedure (actual value) | 23.4 [21 to 27] | 22.1 [12 to 27]
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure): number analyzed (Participants) | 17 | 10
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure) | -0.7 [-2 to 2] | 1.1 [-2 to 10]
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure): number analyzed (Participants) | 17 | 10
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure) | -1.1 [-3 to 1] | 1.5 [-7 to 10]
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure): number analyzed (Participants) | 17 | 10
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure) | -0.5 [-4 to 4] | 0.6 [-3 to 10]
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure): number analyzed (Participants) | 15 | 9
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure) | -0.9 [-4 to 5] | 1.2 [-3 to 10]
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure): number analyzed (Participants) | 17 | 9
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure) | -1.1 [-5 to 5] | 0.8 [-5 to 8]

22. Secondary Outcome: Efficacy: Blood Analysis Parameter -- Base Excess
Description: The blood base excess at all timepoints and the changes from pre-procedure to each timepoint are presented.
  Base excess is defined as the amount of acid that must be added to each litre of fully oxygenated blood to return the pH to 7.40 at a temperature of 37°C and a pCO2 of 40 mmHg (5.3 kPa). The value is reported as a concentration in units of milliequivalent per liter (mEq/L), with positive numbers indicating an excess of base and negative a deficit.
Time Frame: First 72 hours of life (1h, 6h, 24h, 48h, 72h)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mEq/L
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
mEq/L
  Pre-procedure (actual value): number analyzed (Participants) | 18 | 11
  Pre-procedure (actual value) | -3.20 [-6.5 to 1.3] | -5.22 [-15.6 to 3.0]
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure): number analyzed (Participants) | 17 | 10
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure) | -0.49 [-2.5 to 1.7] | 1.07 [-3.0 to 11.1]
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure): number analyzed (Participants) | 17 | 10
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure) | -0.10 [-2.4 to 2.1] | 1.61 [-5.0 to 10.9]
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure): number analyzed (Participants) | 17 | 10
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure) | 0.16 [-2.7 to 3.1] | 2.17 [-5.0 to 15.9]
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure): number analyzed (Participants) | 16 | 8
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure) | -0.29 [-3.8 to 2.6] | 3.21 [-2.0 to 13.2]
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure): number analyzed (Participants) | 17 | 9
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure) | -0.97 [-5.1 to 4.0] | 2.37 [-4.0 to 10.7]

23. Secondary Outcome: Efficacy: Blood Analysis Parameter -- Lactate
Description: The blood concentration of lactate at all timepoints and the changes from pre-procedure to each timepoint are presented.
Time Frame: First 72 hours of life (1h, 6h, 24h, 48h, 72h)
Population: Intention-to-treat population (ITT): All randomized neonates who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
Number analyzed (Participants) | 19 | 12
mmol/L
  Pre-procedure (actual value): number analyzed (Participants) | 11 | 6
  Pre-procedure (actual value) | 2.047 [1.16 to 3.38] | 2.825 [0.60 to 10.50]
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure): number analyzed (Participants) | 9 | 6
  1 h - post procedure (Change from pre-procedure to 1 hour post-procedure) | 0.311 [-0.20 to 1.28] | -0.188 [-1.40 to 0.60]
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure): number analyzed (Participants) | 8 | 6
  6 h - post procedure (Change from pre-procedure to 6 hour post-procedure) | 0.425 [-0.50 to 1.03] | -0.802 [-7.60 to 1.09]
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure): number analyzed (Participants) | 9 | 6
  24 h - post procedure (Change from pre-procedure to 24 hour post-procedure) | 0.009 [-0.30 to 0.56] | -1.100 [-8.50 to 0.70]
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure): number analyzed (Participants) | 9 | 4
  48 h - post procedure (Change from pre-procedure to 48 hour post-procedure) | -0.284 [-1.40 to 1.20] | -2.168 [-8.30 to 0.50]
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure): number analyzed (Participants) | 9 | 5
  72 h - post procedure (Change from pre-procedure to 72 hour post-procedure) | -0.418 [-1.77 to 0.70] | -1.656 [-8.10 to 0.50]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs (SAEs) that started on or after the date of first randomized treatment administration up to the end of the main phase of the study. The main phase of the study included all time points from the pre-randomization period up to and including the follow-up visit at discharge home or 40 weeks PMA, whichever came first.
Description: An AE: defined as "any untoward medical occurrence in a neonate or clinical trial neonate who received the study drug and which did not necessarily have a causal relationship with this treatment", whether or not considered related to the investigational product.
  Safety population (SAF) was used for the analysis of safety. SAF: all randomized neonates who received at least one dose of study treatment.
Arm/Group | Curosurf LISA | Curosurf Endotracheal Tube
All-Cause Mortality (participants affected / at risk) | 1/19 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/12
Other Adverse Events (participants affected / at risk) | 19/19 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curosurf LISA (N=19) | Curosurf Endotracheal Tube (N=12)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curosurf LISA (N=19) | Curosurf Endotracheal Tube (N=12)
Anaemia neonatal (Blood and lymphatic system disorders) | 10 (10) | 4 (4)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Bradycardia neonatal (Cardiac disorders) | 7 (8) | 1 (1)
Neonatal tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Patent ductus arteriosus (Cardiac disorders) | 6 (6) | 5 (5)
Retinopathy of prematurity (Eye disorders) | 7 (7) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema neonatal (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 11 (11) | 5 (5)
Neonatal cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Periumbilical abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 2 (3)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection neonatal (Infections and infestations) | 3 (4) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neonatal hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Poor feeding infant (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 4 (5) | 1 (1)
Periventricular leukomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (4)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypertension neonatal (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor issued an early notification of an immediate enrolment hold to participating study sites (01 June 2022) and an official notification (05 July 2022) after identifying uncertain availability of the CHF 6440 catheter. Because the availability of CHF 6440 catheter to all participating study sites could not be assured, the Sponsor decided to terminate the study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT02772081/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02772081/SAP_001.pdf